CLINICAL TRIAL: NCT03827902
Title: Remote Glycemic Management for Patients With Diabetic Foot Ulcer and Wound Infection
Brief Title: Diabetic Foot Ulcer and Wound Infection
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit participants
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Uma Gunasekaran, Assistant Professor, Internal Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 042018-008
Record Dates: First submitted 2019-01-17; First posted 2019-02-04 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Complications; Diabetes; Diabetic Foot Ulcer; Wound Infection
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus; Diabetic Foot; Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention Group: A Telcare 2.0 BGM, which is FDA cleared, will be used to upload blood glucose measurements to a cloud server accessible by providers. Intervention group will participate in an integrated care model where they will attend Diabetic Clinic and Foot Wound appointments on the same day.
  Interventions: Device: Telcare 2.0 BGM
- Control Group: Control Group will receive usual care (a non-integrated care model where Diabetes Clinic and Foot Wound appointments are on separate days.) These patients will not receive a blood monitoring glucose device.

INTERVENTIONS:
Device: Telcare 2.0 BGM — Blood glucose meter that uploads blood glucose measurements to a cloud server that providers can access and use to monitor patients' glycemic trends.
  Groups: Intervention Group

SUMMARY:
The goal of the study is to compare whether an integrated model of care between Foot Wound and Diabetes Clinic with use of remote glucose monitoring technology (Intervention Arm), as compared with usual care without the use of remote glucose monitoring technology (Control Arm), will result in 1) improved glycemic control, 2) improved ulcer and wound healing, 3) improved patient reported outcomes (PROs), 4) reduced long-term healthcare resource utilization, and 5) improved adherence to anti-glycemic therapy for patients with DFUWI and poor glycemic control over the course of a 6-month intervention period.

DETAILED DESCRIPTION:
This is a two-arm non-randomized convenient pilot trial to assess impact of an active glycemic management model through remote glucose monitoring technology amongst patients with DFUWI and poor glycemic control at the Parkland Diabetes Foot & Wound clinic. The plan is to implement a remote glucose monitoring technology to facilitate improved glycemic management and control. A cellular enabled glucose meter that will upload blood glucose measurements to a cloud server accessible by providers who can remotely review glycemic trends and remotely provide patients with proactive recommendations for treatment adjustments will be used. Patients receiving services in the integrated care model (same day visits in the Foot Wound and Diabetes Clinics at Parkland) will be eligible for inclusion in the intervention arm which includes proactive glucose monitoring guided by remote glucose monitoring technology. Patients receiving usual care services (non-integrated care model clinic days where Foot Wound and Diabetes Clinic visits are on separate days) will be eligible for inclusion in the control arm. The expectation is that patients in the intervention arm will experience greater improvements in glycemic control, compared to the usual care model. The hypothesis is that improved glycemic control in these patients will result in faster healing of diabetic foot wound, infections or ulcers. The effectiveness of the technologically facilitated integrated model of care will be evaluated compared to the usual care using metrics for diabetic foot ulcers and wound healing, glycemic control, patient reported outcomes, health resource utilization and medication adherence after 6 months of intervention. The Telcare 2.0 BGM for remote self-blood glucose monitoring(FDA Cleared) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* 18 years and older
* A1C greater than or equal to 8.5% within the preceding 6 months
* A1C greater than 8% on day of enrollment
* Active diabetic foot ulcer or wound receiving treatment in the Foot Wound clinic at Parkland (ulcer that meets University of Texas Classification Grade 1 or 2 of any stage)

Exclusion Criteria:

* Chronic osteomyelitis (even if completed active therapy)
* Moderate/severe lower limb infection (per Infectious Diseases Society of America criteria)
* Diabetic Foot Ulcer and Wound Infection on Charcot Foot
* Any serious/unstable medical condition that interferes with treatment assignment
* Ankle Brachial Index less than 0.7 or toe pressures less than 30mmHg
* Unwilling to participate or receive injectable treatment or unable to keep appointments
* Non-English or Non-Spanish speakers
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic foot ulcer &/or wound infection and poor glycemic control (A1C ≥ 8.5%) seen in the Foot Wound clinic at a public hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  Mean change in HbA1c from baseline to end of treatment

SECONDARY OUTCOMES:
Glycemic control | 6 months
  Proportion of patients with lower A1C and insulin use
Foot ulcer and/or wound healing | 6 months
  Complete wound healing as defined by University of Texas Health System
Patient reported satisfaction with diabetes treatment | 6 months
  Self-reported outcome assessment questionnaire using the Diabetes Treatment Satisfcation Questionnaire (DTSQ) [Scale range 0-48]; lower scores represent worse outcomes
Patient reported health status | 6 months
  Self-reported outcome assessment questionnaires using the 5 level EQ-5D health status measure (EQ-5D-5L) [Scale range 5-25]; higher scores represent worse outcome
Proportion of patients with emergency department visits | 6 months
  Proportion of patients with emergency department visits following enrollment
Proportion of days covered score | 6 months
  Proportion of days covered score represents an indirect measure of medication adherence and represents the proportion of days medication was dispensed (numerator) over the total potential days the medication should have been dispensed (denominator)
Proportion of patients with hospitalization | 6 months
  Proportion of patients with hospitalization following enrollment
Frequency of invasive procedures | 6 months
  Total number and type of invasive procedures related to diabetic foot ulcer and or wound infection
Number of outpatient visits | 6 months
  Total number of outpatient visits for general or specialized care (including virtual visits) during trial
Number of casts and boots used for treatment | 6 months
  Total number of casts and boots used for treatment related to diabetic foot ulcer and or wound infection
Overall hospital incurred patient-specific cost | 6 months
  Cost (in US $) of overall patient care for Parkland during study enrollment
Cost of glycemic management during study | 6 months
  • Cost of glycemic management during trial, including cost of encounters (including telephone and virtual visits), testing supplies, drug costs, technology costs specifically related to glycemic management

OTHER OUTCOMES:
Frequency of hypoglycemic events | 6 months
  Comparison of frequency of severe hypoglycemic symptoms for usual care versus intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Uma Gunasekaran, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No